CLINICAL TRIAL: NCT04329130
Title: Chidamide Combination With Lenalidomide in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma: an Open Label, Single Arm, Phase II Study
Brief Title: Chidamide Combination With Lenalidomide in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-013
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined Lenalidomide (Experimental): Chidamide, 20 mg, twice per week; lenalidomide, 25 mg, d1-21, and rest for 7 days.
  one treatment cycle per 28 days.For patients with limited lesions and good drug response, local radiotherapy may be assessed by the investigator.
  Interventions: Drug: Chidamide, Lenalidomide

INTERVENTIONS:
Drug: Chidamide, Lenalidomide — All patients enrolled in the study will accept Chidamide combination with lenalidomide regimen.

SUMMARY:
The purpose of this open label,single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of Chidamide combination with lenalidomide for relapsed or refractory peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Histone deacetylase(HDAC) inhibitor has been used in relapsed or refractory peripheral T-cell lymphoma.There are no international studies of Chidamide combination with lenalidomide for relapsed or refractory peripheral T-cell lymphoma. Therefore, this study intends to select the oral HDAC inhibitor Chidamide combined with lenalidomide for relapsed or refractory peripheral T-cell lymphoma, and explore its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* peripheral T cell lymphoma (PTCL);
* no remission or relapse after at least one previous systemic treatment；
* at least one assessable lesion；
* 18-75 years;
* ECOG PS 0-2;
* proper functioning of the major organs;
* expected survival time ≥3 months.

Exclusion Criteria:

* previous received treatment of HDAC inhibitor or lenalidomide;
* central nervous system (CNS) involvement;
* serious heart problems;
* known allergies to experimental drug ingredients;
* diagnosed with or receiving treatment for a malignancy other than lymphoma;
* uncontrolled active infection, with the exception of tumor-related b-symptom fever;
* unable or unwilling to receive antithrombotic therapy;
* history of deep vein thrombosis (DVT) or pulmonary embolism (PE) in the past 12 months;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-03-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
ORR | 4-years
  Overall Response Rate

SECONDARY OUTCOMES:
PFS | 4-years
  Progression Free Survival
DOR | 4-years
  Duration of Overall Response
OS | 4-years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China